CLINICAL TRIAL: NCT06381388
Title: Interaction Between the Brain Hemispheres - Key to Motor Recovery After Stroke
Acronym: InterAct
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jord Vink (Other)
Responsible Party: Sponsor-Investigator, Jord Vink, Coordinating investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL86587.041.24
Record Dates: First submitted 2024-03-17; First posted 2024-04-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Stroke; Transcranial magnetic stimulation; Continuous theta burst stimulation; Upper limb recovery; TMS; cTBS; Interhemispheric inhibition
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active cTBS (Experimental): cTBS delivered with an active TMS coil
  Interventions: Device: cTBS

INTERVENTIONS:
Device: cTBS — A single cTBS session delivered to the contralesional primary motor cortex.

SUMMARY:
Rationale: Acute stroke leaves many patients with functional deficits, of which upper extremity motor impairment is one of the most disabling. Evidence from imaging and electrophysiological studies converge on the idea that impaired motor function after stroke is associated with disrupted network activity in the brain. Non-invasive brain stimulation methods, like transcranial magnetic stimulation (TMS), can be used to restore disrupted network activity and have been shown to successfully facilitate recovery of motor function in patients with stroke. Application of continuous theta burst stimulation (cTBS), an inhibitory form of TMS, to the contralesional motor cortex has been shown to improve the recovery of motor function in patients with stroke. However, responsiveness to this treatment varies considerably between stroke patients and the mechanisms through which contralesional cTBS facilitates recovery of motor function remain unclear.

Objective: To determine if contralesional cTBS normalizes interhemispheric inhibition from the contralesional to ipsilesional primary motor cortex stroke patients with motor impairments. Age-matched healthy persons will serve as controls.

Study design: A prospective, open-label within-subject intervention study

Study population: 40 patients with first-ever ischemic stroke in one hemisphere and a unilateral paresis of the upper extremity, and 40 age-matched controls.

Main endpoints: Primary endpoint: Interhemispheric inhibition from the contralesional to ipsilesional primary motor cortex. Secondary endpoints: contralesional intracortical inhibition; effect of contralesional TMS interference on finger tapping frequency.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age ≥ 18 years;
* First-ever ischemic stroke or intracerebral hemorrhage in a cerebral hemisphere or the brainstem;
* Unilateral paresis of an upper extremity with a Motricity Index (MI) between 9 and 99
* Inclusion possible between 3 weeks and 6 weeks after stroke onset;
* Signed informed consent.

Inclusion Criteria for healthy controls:

* Age ≥ 18 years;
* Signed informed consent.
* Normal motor function with a minimum Motricity Index (MI) of 99.

Exclusion Criteria:

* Disabling medical conditions (severe heart disease, severe head trauma, severe mental illness);
* Severe deficits in communication, memory or understanding which could impede participation, as determined by the treating physician;
* Contraindications to TMS and/or MRI (ferrous implants, history of epilepsy, drug or alcohol abuse over a period of 6 months prior to the experiment, pregnancy);
* Life expectancy shorter than one year;
* Upper limb paresis prior to stroke onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Interhemispheric inhibition (IHI) | Within 30 minutes after cTBS
  Contralesional to ipsilesional IHI measured with a condition pulse delivered over the contralesional M1 and a test pulse delivered over the ipsilesional M1 with an interstimulus interval of 10ms. An aggregated measure (unitless) is obtained by dividing the conditioned motor-evoked potential (MEP) amplitude (in Volts) by the unconditioned MEP amplitude (in Volts). A value smaller than 1 indicates inhibition.

SECONDARY OUTCOMES:
Ipsilesional resting motor threshold (RMT) | Within 30 minutes after cTBS
  Ipsilesional RMT in percentage of machine output. Outcome ranges from 0 to 100%.
Contralesional resting motor threshold (RMT) | Within 30 minutes after cTBS
  Contralesional RMT in percentage of machine output. Outcome ranges from 0 to 100%.
TMS interference | Within 30 minutes after cTBS
  Finger tapping frequency change in response to TMS interference of the contralesional M1.
Intracortical inhibition (ICI) | Within 30 minutes after cTBS
  Intracortical inhibition in the contralesional M1 with an interstimulus interval of 2ms. An aggregated measure (unitless) is obtained by dividing the conditioned motor-evoked potential (MEP) amplitude (in Volts) by the unconditioned MEP amplitude (in Volts). A value smaller than 1 indicates inhibition.

CONTACTS AND LOCATIONS:
Locations (1):
- De Hoogstraat Revalidatie, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No